CLINICAL TRIAL: NCT03990311
Title: Prepared Meals to Prime and Perpetuate Reduced Dietary Sodium Intake in Hemodialysis
Acronym: PEPPERDISH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 999
Record Dates: First submitted 2019-02-04; First posted 2019-06-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Hypertension in Dialysis Patients; Fluid Overload in Dialysis Patients
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: BP, weight, IDH (as defined by an intra-or post dialysis BP <90 mmHg) will be recorded per usual clinical care by the dialysis unit staff.
  Patients will be blinded to the salinity of the salt solutions used to test taste perception and preference.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The experimental arm receives 2 months of sodium restricted prepared meals plus dietary counseling followed by 3 months of counseling alone.
  Interventions: Other: Sodium Restricted Meals
- Control (Placebo Comparator): The control arm receives 5 months of usual care followed by 2 months of receipt of sodium restricted prepared meals.
  Interventions: Other: Control

INTERVENTIONS:
Other: Sodium Restricted Meals — 2 meals prepared with 2 g /day sodium restriction and adhering to dietary recommendations for a hemodialysis patients (phosphate and potassium restricted/ high protein content) 2 meals per day for first month of meal provision period followed by 1 meal per month in the second meal of meal provision period
  Other Names: Dietary Counseling
  Arms: Intervention
Other: Control — Usual Care
  Arms: Control

SUMMARY:
This is a randomized clinical trial in which maintenance hemodialysis patients will be provided with salt restricted 'dialysis friendly' meals and compared to a control arm receiving usual care.

DETAILED DESCRIPTION:
Patients randomized to the intervention arm will receive 2 months of meals plus dietary counseling. Counseling will continue for an additional 3 months while the control arm will have 5 months of usual care followed by 2 months of meal provision. Effects on interdialytic weight gain, achievement of target dry weight, intradialytic hypotension episodes, blood pressure, and a volume assessment using lung U/S to assess lung water will be measured. Salt sensitivity will be tested throughout the study. Self reported questionnaires about the burden of adhering to the low salt diet and the level of adherence with it will be completed at baseline and throughout the study. The investigator hypothesizes that the prepared meals with prime patients behavior and may alter salt taste perception and that these effects will be sustained after the prepared meals have stopped.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18
2. Treated with outpatient hemodialysis for >60 days
3. Mean IDWG over the past 30 days >2 kg
4. Speaks and understands English or Chinese
5. Patient has a freezer at home with space to store at least 7 prepared meals
6. Cognitively intact (able to provide informed consent and answer questionnaires)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Interdialytic Weight Gain throughout Length of Study | Every two weeks starting through 5months (intervention arm)/ 7 months (control arm)
  A standard measurement taken for HD patients at each dialysis session to see weight gained between sessions

SECONDARY OUTCOMES:
Rate of Intradialytic Hypotension Episodes throughout Length of Study | Every two weeks starting at baseline and through 5months (Control Arm)/ 7 months (intervention arm)
  Intradialytic Systolic BP <90 mm Hg

OTHER OUTCOMES:
Pre-dialysis Blood Pressure | through 5months (intervention arm)/ 7 months (control arm)
  BP measurement prior to dialysis, taken for HD patients at each session
Salt Taste Perception | through 5months (intervention arm)/ 7 months (control arm)
  Testing salty solution taste perception via sip, swish, and spit and rating saltiness on a general Labeled Magnitude Scale ranging from "Barely Detectable" to "Strongest Imaginable".
Salt Taste Preference | through 5months (intervention arm)/ 7 months (control arm)
  Testing salty solution taste preference via sip, swish, and spit and, in the opinion of the participant, selecting which solution tasted better.
Fluid Overload | through 5months (intervention arm)/ 7 months (control arm)
  As defined by lung U/S at the end of the dialysis treatment
Rate of Achievement of Estimated Dry Weight | through 5months (intervention arm)/ 7 months (control arm)
  Post-weight not greater than EDW by 0.5 kg

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No